CLINICAL TRIAL: NCT01193387
Title: A Trial to Test for Bioequivalence Between Identical NN1250 Formulations, IM1 and IM2, in Healthy Subjects
Brief Title: Comparison of Two Identical NN1250 Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3769; U1111-1115-5279 (Other: WHO); 2010-018908-83 (EudraCT Number)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (M) IM1 (Experimental)
  Interventions: Drug: insulin degludec
- IDeg (M) IM2 (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Each subject will be allocated to 2 single doses of trial product on 2 separate visits: One injection with formulation 1 and and one injection with formulation 2). Injected subcutaneously (under the skin).
  Arms: IDeg (M) IM1
Drug: insulin degludec — Each subject will be allocated to 2 single doses of trial product on 2 separate visits: One injection with formulation 1 and and one injection with formulation 2). Injected subcutaneously (under the skin).
  Arms: IDeg (M) IM2

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate if two identical formulations of NN1250 (insulin degludec, IDeg) have the same level of drug exposure to the body.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, vital signs and electrocardiogram (ECG), as judged by the Investigator
* Body mass index 18.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the Insulin Degludec concentration-time curve | From 0 to 120 hours after single-dose
Maximum observed Insulin Degludec concentration | From 0 to 120 hours after single-dose

SECONDARY OUTCOMES:
Area under the Insulin Degludec concentration-time curve | From 0 to infinity after single-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com